CLINICAL TRIAL: NCT05097248
Title: Camrelizumab Combined With Liposomal Doxorubicin and Losartan in the Treatment With Advanced or Locally Advanced Triple-negative Breast Cancer Who Have Received no More Than 1 Prior Line of Chemotherapy
Brief Title: Camrelizumab in Combination With PLD and Losartan in Patients With TNBC Who Have Received ≦ 1 Line of Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry); CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yanxia Zhao, Director of the Department of Breast Oncology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WHUH-BC-001
Record Dates: First submitted 2021-10-11; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — camrelizumab; liposomal doxorubicin; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab, Liposomal doxorubicin and Losartan (Experimental): Participants receive intravenous camrelizumab (200 mg, Q3W) and liposomal doxorubicin (40 mg, Q3W for 6 weeks) plus oral losartan (50 mg loading dose followed by 100 mg QD, Q3W, until discontinuation of liposomal doxorubicin).
  Interventions: Drug: Camrelizumab; Drug: Liposomal Doxorubicin; Drug: Losartan

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab 200mg (3mg/kg for patient whose weight is below 50kg) will be administered as an intravenous infusion over 30 minutes every three weeks until unacceptable toxic effects or disease progression or other termination criteria appeared.
Drug: Liposomal Doxorubicin — Liposomal Doxorubicin 40 mg/m2 on D1 every 3 weeks; 6 cycles are planned to be completed or discontinued due to intolerable toxicity or progression.
Drug: Losartan — Losartan will be orally administered at 50 mg for three days and increased to 100 mg if tolerated until the whole course of chemotherapy; if not tolerated, it will be maintained at 50 mg until the whole course of chemotherapy

SUMMARY:
This is a phase II, single-arm, multi-center, prospective clinical study of camrelizumab in combination with liposomal doxorubicin and losartan in patients with advanced or locally advanced triple-negative breast cancer who had received no more than 1 prior line of chemotherapy. Our aim was to explore the efficacy and safety of it.

DETAILED DESCRIPTION:
This a phase II, open-labeled, multi-centered, single-arm, investigator-initiated clinical trial to assess the efficacy and safety of camrelizumab combination with liposomal doxorubicin and losartan in female patients age of 18 to 70 with advanced or locally advanced TNBC, and previously treated with no more than one line of chemotherapy in the advanced setting. The number of patients to be included is 52 patients (Simons two stage design). All enrolled patients will be treated with camrelizumab 200mg (iv. 3mg/kg for patient whose weight is below 50kg) on day 1 of each 21-day cycle, and liposomal doxorubicin (40 mg, Q3W for 6 weeks) plus oral losartan (50 mg loading dose followed by 100 mg QD, Q3W, until discontinuation of liposomal doxorubicin).The primary objective is to assess the overall response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-70.
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
3. The pathologic diagnosis of unresectable recurrent or metastatic triple-negative breast cancer ［ER-negative(IHC<1%), PR-negative(IHC<1%), HER2-negative（IHC-/+ or IHC++ and FISH/CISH-）］. Patients with at least one measuring lesion that was conformed to RECIST v1.1 standard.
4. With a life expectancy of at least 12 weeks.
5. The cumulative dose of prior doxorubicin and epirubicin should not exceed 300 mg/m2 and 600 mg/m2, respectively, with randomization > = 12 months since last treatment.
6. Previously treated with no more than one line of chemotherapy in the advanced setting.
7. PD-L1 positive, CPS score ≥ 1.
8. At least one measurable lesion according to RECIST 1.1;
9. The functional level of major organs must meet the following requirements:

   1. blood routine: neutrophil (ANC)≥1.5×10^9/L; platelet count (PLT)≥90×10^9/L; hemoglobin (Hb) ≥90 g/L;
   2. blood biochemistry: total bilirubin (TBIL)≤upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5×ULN; alkaline phosphatase ≤ 2.5×ULN; blood urea nitrogen (BUN) and creatinine (Cr)≤1.5×ULN;
   3. coagulation: international normalized ratio (INR) or prothrombin time (PT)≤1.5×ULN; activated partial thromboplastin time (APTT) ≤1.5×ULN.
   4. Heart: left ventricular ejection fraction (LVEF)≥50% as assessed by echocardiography (ECHO) or multigated acquisition (MUGA).
   5. Thyroid function: thyroid stimulating hormone (TSH) ≤ ULN; if abnormal, T3 and T4 levels should be investigated, and normal T3 and T4 levels can be included.
10. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose and must be willing to use very efficient barrier methods of contraception for the course of the study through 6 months after the last dose of study treatment.
11. The patient can swallow pills.
12. The patients sign the written informed consent.

Exclusion Criteria:

1. The subjects had a central nervous system metastases with clinical symptoms.
2. Other clinical trials of drugs were used in the first four weeks before the first dose.
3. Subjects with severe allergic reactions to other monoclonal antibodies.
4. Received other anti-tumor treatments within 28 days before the first dose.
5. A heart condition or disease that is not well controlled.
6. Subjects with treatment history of anti-angiogenesis drugs, or immunotherapy (previous use of anti-PD-1/PD-L1 antibodies was allowed) or eribulin.
7. The subjects had any history of autoimmune disease or any use of systemic glucocorticoid or immunosuppressive medications.
8. Subjects had history of hypertension and poor control with antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥100 mmHg)；
9. Subjects must not have baseline hypotension, defined as systolic blood pressure less than 100 mmHg in both readings taken 2 days prior to the study.
10. Urine routine indicated that urine protein ≥ ++, or the 24-hour urine protein quantity ≥ 1.0g.
11. Hereditary or acquired bleeding and thrombotic tendencies (such as hemophilia, coagulation dysfunction, thrombocytopenia, hypersplenism, etc.).
12. Human immunodeficiency virus (HIV) infection, active hepatitis B (hepatitis B indicates antigen positive and HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody positive and HCV-RNA above the lower limit of detection of the analytical method).
13. Receive live vaccine within 4 weeks before or during the study period;
14. Patients who are allergic to or contraindicated to the experimental drugs.
15. Concurrent medical conditions that, in the judgment of the investigator, would jeopardize the subject's safety, could confound the study results, or affect the subject's completion of this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Estimated 12 months
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Estimated 12 months
  PFS was defined as the time from randomization to first documented disease progression (PD) using Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) or death from any cause, whichever occurred first. For target lesions, PD was defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since treatment started or the appearance of 1 or more new lesions. For non-target lesions, PD was defined as the appearance of 1 or more new lesions and/or unequivocal progression of existing non-target lesions.
Overall Survival (OS) | Estimated 24 months
  Overall Survival (OS), defined as the time from the date of randomization to the date of death, regardless of the cause of death. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last study medication and participants with no post-baseline information were censored at the date of randomization.
Duration of Response (DoR) | Estimated 12 months
  DoR is defined as date of initial confirmed PR/CR until date of progressive disease or death from any cause. PR or CR or SD is according to RECIST version 1.1.
Clinical Benefit rate (CBR) | Estimated 12 months
  Ratio of CR,PR and SD greater than or equal to 24 weeks in all subjects
Adverse events (AEs) | Estimated 12 months
  AEs were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0.3.
  In general, AEs are graded according to the following: Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE.
  The type, grade and frequency of AEs will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Zhao, M.D., Study Chair — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College of HUST, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No